CLINICAL TRIAL: NCT00558493
Title: Phase lV Study to Evaluate the Safety and Effectiveness of Switching Treatment From Lamivudine to Clevudine in the Chronic Hepatitis B Patients With Suboptimal Virologic Response During Lamivudine Treatment
Brief Title: Switching Study From Lamivudine to Clevudine in the Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-406; KB-406
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — clevudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): switching treatment from lamivudine to clevudine
  Interventions: Drug: Clevudine

INTERVENTIONS:
Drug: Clevudine — clevudine 30 mg qd for 24 seeks

SUMMARY:
A multi-center and open study to compare the safety and effectiveness of switching treatment from lamivudine to clevudine for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HBV DNA > 2,000 copies/mL at screening
* Patients who have compensated liver disease (Child-Pugh score =<6)
* Patients without LMV resistant mutation by RFMP assay
* Patients who have NOT experienced viral breakthrough at consecutive two measurements (at least one month apart) during lamivudine monotherapy
* Patients who can submit the written consent and comply with the claims postulated of this clinical trial

Exclusion Criteria:

* Currently receiving antiviral except LMV or corticosteroid therapy
* Patients that previously received antiviral treatment for hepatitis B other than lamivudine in the proceeding 12 months
* Previous treatment with interferon or other immunomodulatory therapies must have ended at least 6 months preceding the study screening
* Treatment with nephrotoxic drugs, competitors of renal excretion, and/or hepatotoxic drugs within 2 months before study screening or during the study period
* Patients who is co-infected with HCV, HDV or HIV
* Serious concurrent medical conditions
* Prior organ transplantation
* Patient has creatinine clearance less than 60mL/min as estimated by the following formula:

[(140-age in years) (body weight [kg])] / [(72) (serum creatinine] [mg/dL])[Note: multiply estimates by 0.85 for women]

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-11

CONTACTS AND LOCATIONS:
Locations (1):
- Youngnam University Medical Center, Daegu, South Korea